## Title: Ultrasound Guided Local Infiltration Analgesia for Hip Arthroscopy

PI: Sanjay K. Sinha, MD

NCT01907191

Document Date: June 11, 2013

## Ultrasound Guided Local Infiltration Analgesia for Hip Arthroscopy Protocol

Sanjay K. Sinha, MD
Department of Anesthesiology
Saint Francis Hospital and Medical Center
114 Woodland Street, Hartford, CT 06105

### **Table of Contents:**

## **Study Schema**

- 1.0 Background
- 2.0 Rationale and Specific Aims
- 3.0 Inclusion/ Exclusion Criteria
- 4.0 Enrollment
- 5.0 Study Procedures
- 6.0 Reporting of Adverse Events or Unanticipated Problems
  Involving Risk to Participants or Others
- 7.0 Study Withdrawal/ Discontinuation
- 8.0 Statistical Considerations
- 9.0 Privacy/ Confidentiality Issues
- 10.0 Follow-up and Record Retention

## 1.0 Background

Patients undergoing hip arthroscopy experience moderate to severe postoperative pain. Effective pain control after surgery is an important component in the overall management of these patients. Good pain control encourages early participation in rehabilitation program, increases success of the surgery, and improves patient satisfaction. Typically, postoperative analgesia is provided to these patients either with nerve blocks (psoas compartment lumbar plexus block and sciatic nerve block) or opioid medications (1,2,3). Both these methods provide good pain relief but nerve blocks are associated with weakness of lower extremity muscles which interferes with early ambulation and increase the risk of falls while narcotic medications increase the risk of nausea, vomiting, itching, constipation, ileus, urinary retention, sedation and respiratory depression.

Liposomal bupivacaine has the same active ingredients as bupivacaine. Both act to block the generation and conduction of nerve impulses associated with pain. Liposomal bupivacaine consists of bupivacaine encapsulated within a hydrophobic lipid membrane. Bupivacaine is released from the multivesicular liposomes over a prolonged period of time. (4)

- Lumber Plexus Blockade Reduces Pain After Hip Arthroscopy: A Prospective Randomized Controlled Trial. YaDeau J, Tedore T, Goytizolo E, Kim D, Green D, Westrick A, Fan R, Rade M, Ranawat A, Coleman S, Kelly B. Anesthesiology & Analgesia 2012; 115(4): 968-972.
- 2. The analgesic impact of preoperative lumbar plexus blocks for hip arthroscopy. A retrospective review. Schroeder K, Donnelly M, Anderson B, Ford M, Keene J. Hip International 2013; 23(1): 93-8.
- 3. Are Femoral Nerve Blocks Effective for Early Postoperative Pain Management After Hip Arthroscopy? Ward J, Albert D, Altman R, Goldstein R, Cuff G, Yourn T. Arthroscopy: The Journal of Arthroscopic and Related Surgery 2012; 28(8): 1064-69.
- 4. Liposomal bupivacaine: A long-acting anesthetic for postsurgical analgesia. Formulary 2012.

## 2.0 Rationale and Specific Aims

Ultrasound guided peri-articular Hip infiltration with local anesthetic solution is an alternative analgesic technique that has been shown to reduce pain, opioid consumption and facilitate earlier discharge from hospital after surgery without causing any weakness of lower extremity. The typical duration of analgesia after peri-articular analgesia lasts only for 8-10 hours. When the effect of injected local anesthetic solution wears off, patients start relying on opioid pain medications for pain control. By using long acting liposomal bupivacaine for LIA we hypothesized that we will provide prolonged duration of analgesia and significantly reduce pain tablet consumption.

#### 3.0 Inclusion/Exclusion Criteria

Inclusion Criteria:

- 1. Patients having hip arthroscopy
- 2. Patients between the ages of 18-80 years

#### **Exclusion Criteria**

- 1. History of neurologic disease, neuropathy, diabetes
- 2. Allergy to local anesthetic solution
- 3. Chronic use of narcotics
- 4. History of previous hip arthroscopy on the ipsilateral side
- 5. Pregnancy

#### 4.0 Enrollment

Subjects will be consented in a private area prior to surgery. An investigator will explain the study and answer all questions.

## 5.0 Study Procedures

1. Preoperative evaluation and consent

2. General anesthesia for hip arthroscopy

3. Ultrasound guided injection of liposomal bupivacaine (experimental group) or bupivacaine (control group) (around the anterior, lateral and medial aspect of hip joint.

4. Hip arthroscopy

5. Postoperative recovery – assessment of pain and narcotic consumption using pain scores and 14-question survey

6. Discharge of patients from hospital to home

7. Patient records pain scores and completes 14-question survey

8. Follow up by telephone 24 hours and 96 hours after surgery to collect data

# 6.0 Reporting of Adverse Events or Unanticipated Problems Involving Risk to Participants or Others

If there are adverse events or unanticipated problems involving risk to the participants or others, they will be reported to the IRB within five working days after their occurrence.

## 7.0 Study Withdrawal/ Discontinuation

If the participant requests to be withdrawn from the study, the investigator will inform participant that their standard of care will remain the same and that there are no adverse indications from withdrawing. Their withdrawal statement will be added to the participant's Consent Form. The corresponding Study Subject Number will be removed from the study list. Discontinued participant records will not be used to compile the final report.

#### 8.0 Statistical Considerations

S 5

Continuous data will be analyzed using parametric methods for normal distribution and non-parametric methods for non-normal distribution (Student t-test or Mann Whitney/Wilcoxon Sum test). Chi-squared or Fisher's exact tests will be used to analyze categorical data. Statistical significance will be set at  $\alpha < 0.05$ 

Sample size of 36 was calculated based on our assumption that a mean difference of 1.0mg ( $\pm 1$  SD) in intravenous hydromorphone administration in the recovery room between the experimental group and control group with a power of 80 % and  $\alpha = 0.05$  (2 sided test) and a 10% dropout. Included is the power analysis:

```
t tests - Means: Difference between two independent means (two groups) Analysis: A priori: Compute required sample size Input: Tail(s) = Two Effect size d = 1.0  
\alpha err prob = 0.05  
Power (1-\beta err prob) = 0.80  
Allocation ratio N2/N1 = 1  

Output: Noncentrality parameter \delta = 2.9154759  
Critical t = 2.0369333  
Df = 32  
Sample size group 1 = 17  
Sample size group 2 = 17  
Total sample size = 34  
Actual power = 0.8070367
```

## 9.0 Privacy/ Confidentiality Issues

Patients will be assigned a study subject number that will be used on all data collection documents. Their personal information (Name, address, telephone number, age, weight, height, sex, etc.) will only be recorded on one list with study subject numbers. This list will be separate from all other documents under lock and key and only used to make follow up phone calls. Study records are kept confidential. If the results of the study are published in a scientific journal or presented at a scientific meeting, the subjects' names and any identifiers will not be used.

## 10.0 Follow-up and Record Retention

The duration of the study will last 96 hours after the participant's total knee replacement. Study records will be stored for three years after the close of the study. Study records will then be destroyed using the standard Saint Francis shredding service.



## SAINT FRANCIS HOSPTIAL AND MEDICAL CENTE

Institutional Review Board
Full Board Application for Initial Project Approval



All applications must be typed. Point, click and type in the appropriate cell; cells will expand to accommodate text. Tabbing out of the last cell on the right of a table will insert another row. Referencing the protocol is not acceptable since not all IRB members receive the complete protocol. The IRB reserves the right to return applications that do not provide sufficient responses.

There are consent form templates available for the following study categories, their use is recommended but not required.

#### Study Categories:

- 1. For investigational studies involving drug or devices, all sections of this application need to be completed. Use consent template 1.
- 2. For Full Board social or behavioral research, sections: 1, 2, 3, 4, 5.0-5.3, 6, 7, 8, 9, 10, 11, and 13 need to be completed. Use consent template 2.
- 3. For establishment of a research registry, sections: 1, 2, 3, 4, 5.0-5.3, 6, 7, 8, 9, 10 and 13 need to be completed. Use consent template 3.

| SECT | ION 1 - BASIC STUDY INFO | DRMATION | | |
|---|---|---|---|---|
| 1.0 | Type of Submission: X Initial Application Resubmission to Address Contingencies | | | |
| 1.1 | Name of Principal Inve | estigator for IRB Proposal | : Sanjay K. Sinha | |
| 1.2 | | Project location: AMERICA CENTER | X SAINT FRANCIS CAMPUS | ☐ BURGDORF CLINIC/BANK OF |
| | | ☐ MOUNT SINAI CAMPUS ☐ OTHER (PLEASE SPECIF | ☐ ASYLUM HILL FAMIL<br>FY): | Y MEDICINE |
| 1.3 | Type of review reques | ted: X FULL BOARD | | |
| 1.5 | Complete Associated | stoperative Analgesia after l | пір Антиосору. | |
| 1.6 | Name of PI on the gra | nt: N/A | | |
| 1.7 | Abbreviated Project T | itle: Ultrasound Guided Lo | ocal Infiltration Analgesia fo | r Hip Arthroscopy |
| 1.8 | Identify any external f | unding source for this stu | ıdy: N/A | |
| 1.9<br>Anes | | unding source for this stu<br>lospital and Medical Center | dy (e.g. Academic Affairs, dept. fund<br>, Hartford, CT. | is etc.): Department of |
| 1.10 | ldentify the sponsor f | or this study (e.g. PI, ECOG, | Pfizer, etc): N/A | |
| 1.11 | - | | est or other relationship with<br>by each investigator and submitted v | |
| 1.12 | Will the PI benefit per | sonally from this study? | ☐ YES X NO | |
| 1.13 | Will the sponsor inde | mnify subjects in the ever | nt of a research-related injui | y? □ YES X No |

| | | | | Machan M. |
|---|---|---|---|---|
| SECT | ION 2- RESEARCH PERSON | NNEL INFORMATION | | 5/1 8 |
| | | PRINCIPAL INVESTIGATOR (last, first) | STUDY COORDINATOR (last, first if other than PI) | CONTACT PERSON (last, first if other than PI or SC) |
| 2.0 | Name | Sinha, Sanjay | Patricia Gallo | |
| 2.1 | Degree(s) Held | MD | Associates in Science | |
| 2.2 | Professional<br>Licenses (type & #) | MD # 035260 | | |
| 2.3 | Professional<br>Certifications | Board Certification in<br>Anesthesiology | | |
| 2.4 | Job Title | Anesthesiologist | Executive Adm. Assistant To Chief of Staff | |
| 2.5 | Department | Anesthesiology | Anesthesiology | |
| 2.6 | Mail Code | 30301 | 30301 | |
| 2.7 | Phone Number | 860-714-9666 | 860-714-9666 | |
| 2.8 | Emergency Number | 860-714-6654 | 860-830-8629 | |
| 2.9 | Fax Number | 860-714-8110 | 860-714-8419 | |
| 2.10 | Pager Number | 762-1589 | | |
| 2.11 | E-mail Address | sanjaysinha@comcast.net | pgallo@stfranciscare.org | |
| 2.12 | Other Affiliations of<br>PI (e.g. CCMC, Hartford<br>Hospital, Storrs, UCHC) | | ***** | 在在在在在安全的企业会在全有的有关的有关的有效的。 |

2.13 Off-hours/weekend contact information (Optional):

2.14 Provide a brief summary of the qualifications of the PI to conduct this study and attach an NIH biosketch or complete CV. See attached CV

2.15 Provide information on co-investigators for the study (tabbing out of the bottom right cell will insert another row if needed)

| Name<br>(Last, First) | Degrees<br>Held | Licenses<br>(type, St. #) /<br>Certifications | Department | Affiliation | Primary Function(s) Performed In Study |
|---|---|---|---|---|---|
| Jonathan Abrams | MD | MD #024924 | Anesthesiology | SFHMC | Anesthesiologist,<br>design of study,<br>consent, data<br>analysis |
| Sivasenthil Arumugam | MD | MD #044509 | Anesthesiology | SFHMC | Anesthesiologist, Data analysis |
| John D'Alessio | MD | MD #030269 | Anesthesiology | SFHMC | Anesthesiologist, data analysis |
| William Suter | Underg-<br>raduate<br>student,<br>class of<br>2016 | | Summer<br>Research Intern,<br>Department of<br>Anesthesiology | | Design of study,<br>data collection, data<br>entry |

| Additional Information | on on Co-Investig | jators (e.g. previous | s research exper | ience): | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | · | |
| Attach an NIH biosk | etch or comple | ete CV for each | co-investiga | tor. | | | |
| Provide information | on research a | ssistants for the | e study (tabbir | ng out of the bottom ri | ght cell will inser | t another row if I | needed) |
| Name | Degrees | Licenses | Departn | nent Affilia | | Primary Fund | |
| (Last, First) | Held | (type, St. #) /<br>Certifications | | | | Performed Ir | n Study |
| | 1 | Cerufications | | | | | |
| | | - | | | | | |
| Additional Information | on on research a | ceietante (e a prei | vious research e | vnerience): | | | |
| Augmonia mionnau | on research a | ssistants (e.g. pie | vious research e | хрененосу. | | | |
| | | | <u></u> | <u> </u> | <u> </u> | | |
| ECTION 3 - COLLABO | DRATING INSTITUT | TIONS / MULTI-CE | NTER TRIALS | | | | |
| | | ites involved w | ith this stud | y? □YES X | No | | |
| , | If yes, proceed to | ` | Land State | | | | |
| .1 If collaborating | with other sites | s, provide the na | ame of each | institution, and | place an x u | nder the col | lumn(s) |
| that describes to obtained IRB ap | | | | , Provide the da | ite that the o | mer msmu | IOII |
| Optained into ap | provar or maio | ate that it is per | iding. | 10 SEE | | | |
| Institution's Name | Recruitment | | Interactions | Interventions | Follow-up | Analysis | IRB<br>Approva |
| | 8 | Consenting<br>Subjects | (e.g. survey) | (e.g. needle stick) | | 651 | Date |
| tions of a s | A | | | | | = = = | |
| | | TOTAL VENTURE | | | | | |
| Additional Comme | ante: | | | | | | |
| Additional Comme | ints. | | | | | | |
| O Indicate the o | vnootod noroor | tage of enrollm | ont at each | annlicable cite | and place ar | Y in the an | propriate |
| .2 Indicate the e | xpecteu percer<br>e which institu | tion, based on t | he preponde | erance of the ex | pected enrol | Iment, you | are |
| requesting se | rve as the IRB | of record or tha | t independe | nt IRB approval | will be soug | ht from eac | h |
| applicable site | e. | | | | | | |
| Institution's Nar | ne % to be Eı | rolled/Consente | d Reques | ted IRB of Record | Indepe | ndent IRB Re | view |
| SFHMC | 45 1 2. | | | with the second part of the seco | | | |
| | II_ FRESH | PEND TRANSFER | | | MEN MEN | | 1 7 8 |
| nformation on mul | ti-center trials | | | | | | |
| .3 Is this a multi | -center trial? (I | f no, skip to section | n 4, if yes proc | eed to 3.4) | YES X No | | |
| | | | | Hay of A | | | |
| .4 Will SFHMC s | erve as the lea | d institution? | | 3 No | | | |
| | | | | | t madificatio | na unantia | hatad |
| | plans for comn<br>I interim result: | nunication amo | ng sites in to | erms of protoco | i modificatio | ns, unantic | pated |
| hionicilia alio | | | | | | | |
| SECTION 4 - PROJECT | T CHARACTERIST | ICS, SUMMARY AN | ID DESIGN | | | | |
| | | frame during w | | dy will be cond | ucted: | | |
| | 333 W-W-H- | | | | | (44) | / |
| Expected Star | Expected Start Date (mm/dd/yyyy): Expected Completion Date (mm/dd/yyyy): | | | | | | |

| | | heat describe v | our study /o o o | neor gastrointes | inal |
|---|---|---|---|---|---|
| pancreatic or psychiatry, addictive be | eutic area and sub-area(s) that ehaviors, gambling). | best describe y | our study (e.g., ca | micer, gastronites | arrea, |
| Primary Area | Sub- Area | | 2 <sup>na</sup> Sub- Area | | |
| Ambulatory Surgery | Recovery Room | | | | |
| Place an X after the applica | able study phase: | | | | |
| Phase I Phase II | Phase III Phase IV | (Post Marketing | ) X Not a c | linical trial | |
| Thase I I hade it | 11100111 | - II | | | - |
| | | | 1 | af Alaia alaasa | bee |
| For post-marketing trials, of | lescribe any post-marketing re | equirements imp | posed on the use | e of this drug | by |
| the FDA. NONE | | | | | |
| the PDA. NONE | | | | | |
| | | | | 11.5 | _ |
| Place an Y after all charact | eristics that are applicable to t | the study design | n: | | |
| Place all A after all charact | ensues that are approause to | | | S. Day San Land | - |
| Pilot Study | Case-Control | Rand | omization | X | |
| 1 not other | Study | | 100 | | |
| - 10/1 | | Place | ha | 3 - 3 - 3 - 3 - 3 - 3 | |
| Observational Study | Double-blind | | | | $\dashv$ |
| Cross-Sectional Study | Chart review | Norm | al Controls | | |
| Survey | Focus Group | | | | |
| Other (specify): Observer Bl | linded | Strong to the section with | TOWN THE REAL PROPERTY. | | |
| Other (specify). Observer br | IIIded | | | | |
| | | | | 11-11-11-11-11-11-11-11-11-11-11-11-11- | - |
| | | | O I I I I I | | |
| Provide 2 or 3 sentences d | lescribing your project in lay to | erms. We have a | previously shown | that injecting I | oca |
| Floyide 2 of a sentences a | joint under ultrasound guidance | prior to start of s | urgery will decrea | se the pain a | nd |
| sthetic solution around the hip | Joint under ultrasound guidance | prior to start or s | - are the pair cont | trol using eithe | ar. |
| n-medication requirements afte | r surgery. This study is being un | denaken to com | pare the pain con | tioi using citie | 70<br>70 |
| ivacaine versus liposomal bupi | ivacaine. Liposomal bupivacaine | can potentially | provide pain relief | lasting up to | 12 |
| www.bita.com.ulon.bumiumonino.or | an provide pain relief up to 12 ho | ours. | | | |
| re write regular attolyacation ta | an provide paint rener up to 12 to | | | | |
| rs while regular publicacaine ca | | | | | S 1100 |
| | | 4.7, 4.8 and 4.9 com | bined should not exce | ed the equivalent | of fi |
| | ion of this project. (Responses | | | | |
| Provide a summary descript | tion of this project. (Responses | | | TRULE CONST. | 5 |
| Provide a summary descript pages) | | diversión G | | | tion |
| Provide a summary descript pages) | | is to compare the | efficacy and dur | ation of intiltra | |
| Provide a summary descript pages) | ims: The objective of this study i | is to compare the | e efficacy and dur | ation of intiltra<br>bupivacaine f | or L |
| Provide a summary descript pages) /potheses, Objectives and Allegasia between liposomal but | ims: The objective of this study i | ne. By using long | acting liposomal | bupivacaine r | OT L |
| Provide a summary descript pages) /potheses, Objectives and Allegasia between liposomal but | ims: The objective of this study i | ne. By using long | acting liposomal | bupivacaine r | OT L |

Patients undergoing hip arthroscopy experience moderate to severe postoperative pain. Effective pain control after surgery is an important component in the overall management of these patients. Good pain control encourages early participation in rehabilitation program, increases success of the surgery, and improves patient satisfaction. Typically, postoperative analgesia is provided to these patients either with nerve blocks (psoas compartment lumbar plexus block and sciatic nerve block) or opioid medications (1,2,3). Both these methods provide good pain relief but nerve blocks are associated with weakness of lower extremity muscles which interferes with early ambulation and increase the risk of falls while narcotic medications increase the risk of nausea, vomiting, itching, constipation, ileus, urinary retention,

sedation and respiratory depression.

Ultrasound guided peri-articular Hip infiltration with local anesthetic solution is an alternative analgesic technique that has been shown to reduce pain, opioid consumption and facilitate earlier discharge from hospital after surgery without causing any weakness of lower extremity. The typical duration of analgesia after peri-articular analgesia lasts only for 8-10 hours. When the effect of injected local anesthetic solution wears off, patients start relying on opioid pain medications for pain control. By using long acting liposomal bupivacaine for LIA we hypothesized that we will provide prolonged duration of analgesia and significantly reduce pain tablet consumption.

Liposomal bupivacaine has the same active ingredients as bupivacaine. Both act to block the generation and conduction of nerve impulses associated with pain. Liposomal bupivacaine consists of bupivacaine encapsulated within

a hydrophobic lipid membrane. The lipid membrane forms numerous capsules of the drug that are independent of each other (liposomes). Bupivacaine is released from the multivesicular liposomes over a prolonged period of time. (4)

- Lumber Plexus Blockade Reduces Pain After Hip Arthroscopy: A Prospective Randomized Controlled Trial. YaDeau J, Tedore T, Goytizolo E, Kim D, Green D, Westrick A, Fan R, Rade M, Ranawat A, Coleman S, Kelly B. Anesthesiology & Analgesia 2012; 115(4): 968-972.
- 2. The analgesic impact of preoperative lumbar plexus blocks for hip arthroscopy. A retrospective review. Schroeder K, Donnelly M, Anderson B, Ford M, Keene J. Hip International 2013; 23(1): 93-8.
- Are Femoral Nerve Blocks Effective for Early Postoperative Pain Management After Hip Arthroscopy? Ward J, Albert D, Altman R, Goldstein R, Cuff G, Youm T. Arthroscopy: The Journal of Arthroscopic and Related Surgery 2012; 28(8): 1064-69.
- 4. Liposomal bupivacaine: A long-acting anesthetic for postsurgical analgesia. Formulary 2012.

#### **Preliminary Studies:**

Please attach a copy of the full protocol if available.

- 4.7 Provide an outline of the experimental design addressing the following: time line of the study from initiation through data analysis, procedures including a time sequence of when those procedures that involve human subjects will be performed and how they will be monitored.
  - 1. Preoperative evaluation and consent
  - 2. General anesthesia for hip arthroscopy
  - 3. Ultrasound guided injection of liposomal bupivacaine (experimental group) or bupivacaine (control group) (around the anterior, lateral and medial aspect of hip joint.
  - 4. Hip arthroscopy
  - 5. Postoperative recovery assessment of pain and narcotic consumption
  - 6. Discharge of patients from hospital to home
  - 7. Follow up by telephone 24 hours and 96 hours after surgery

#### Description of sample size:

Two groups of 18 patients each.

Estimated enrollment per year: All subjects will be enrolled in a year

#### Primary and secondary outcomes and endpoints:

Primary outcome measures will be opioid consumption. Opioid consumption will be recorded intraoperatively (during the surgery), in recovery room and at home after discharge from hospital. Secondary outcome measures will be pain scores (at rest and ambulation) sleep disturbances, constipation, nausea/vomiting and satisfaction with pain management.

4.8 Describe methods of analysis, sample size supported by appropriate power calculations.

Continuous data will be analyzed using parametric methods for normal distribution and non-parametric methods for non-normal distribution (Student t-test or Mann Whitney/Wilcoxon Sum test). Chi-squared or Fisher's exact tests will be used to analyze categorical data. Statistical significance will be set at  $\alpha < 0.05$ 

Sample size of 36 was calculated based on our assumption that a mean difference of 1.0mg ( $\pm 1$  SD) in intravenous hydromorphone administration in the recovery room between the experimental group and control group with a power of 80 % and  $\alpha$  = 0.05 (2 sided test) and a 10% dropout. Included is the power analysis :

t tests - Means: Difference between two independent means (two groups)

Analysis: A priori: Compute required sample size

Input:

Tail(s) = Two

Effect size d = 1.0

 $\alpha \, \text{err prob} = 0.05$ 

Power (1- $\beta$  err prob) = 0.80

Allocation ratio N2/N1 = 1

Output: Noncentrality parameter  $\delta = 2.9154759$ 

Critical t = 2.0369333

Df = 32

Sample size group 1 = 17

Sample size group 2 = 17

Total sample size = 34

Actual power = 0.8070367

4.9 List specific clinical eligibility requirements for subjects, and clinical criteria that would exclude otherwise acceptable subjects.

| _ | Inclusion Criteria | Exclusion Criteria |
|---|---|---|
| a. | Patients having Hip Arthroscopy | History of neurologic disease, neuropathy, diabetes |
| b. | Age 18 – 80 years | Allergy to local anesthetic solution |
| C. | The state of the s | Chronic use of narcotics |
| d. | | Inability to give consent/cooperate with study |
| e. | | History of previous hip arthroscopy on the ipsilateral side. |
| _ | | Pregnancy |

4.10 Provide the age range or age description of subjects and justification for the age selection:

18 - 80 years

4.11 Are there any non-clinical factors that will exclude subjects, e.g. race/ethnicity, gender, language? If so, justify why the exclusion is necessary. Only English speaking subjects will be included in the study to ensure that the patients understand the protocol, give informed consent and cooperate with the study

SECTION 5 -PROTECTION AGAINST AND MINIMIZATION OF RISKS (45 CFR 46.111(A)(1))

5.0 List all procedures to be performed on human subjects. Also list alternative therapies or procedures that may be advantageous to the subject. Discuss the risks and benefit of any alternative therapy.

Non-Experimental Procedures: Administering oral or intravenous pain medications, Ultrasound guided injection of bupivacaine around hip joint

Experimental Procedures: Ultrasound guided injection of liposomal bupivacaine around the hip joint

Alternative Options: Conventional use of intravenous and oral pain medications; psoas compartment lumbar plexus block; bupivacaine as locally injected anesthetic

**Risks and Benefits of Alternatives:** 

Benefit: will provide adequate postoperative analgesia

Risk: increased risk of nausea vomiting, sedation, respiratory depression, urinary retention

4.9 Describe the potential risks associated with the proposed research, the procedures to protect against or minimize potential risks and assess the likelihood of the risk occurring and if it were to occur the seriousness to the subject.

| Physical Risks: | Procedures to Protect<br>Against / Minimize Risks | Occurrence | Seriousness to Subject if<br>Risk Occurs |
|---|---|---|---|
| 711010101010101010101010101010101010101 | Vital sign monitoring<br>(Continuous EKG, Blood | Rare | Majority of risks are not permanent in nature |

| | anesthetic toxicity -Infection | pressure, pulse oximetry, capnography) emergency drugs readily available, including Intralipid 20% to treat local anesthetic toxicity, use standard sterile precautions and aseptic injection technique to avoid risk of infection | | |
|---|---|---|---|---|
| | Psychological Risks: | Procedures to Protect<br>Against / Minimize Risks | Likelihood of Occurrence | Seriousness to Subject if<br>Risk Occurs |
| | n/a | | | |
| | Economical Risks: | Procedures to Protect<br>Against / Minimize Risks | Likelihood of<br>Occurrence | Seriousness to Subject if<br>Risk Occurs |
| | None | | | |
| | Social Risks: | Procedures to Protect Against / Minimize Risks | Likelihood of Occurrence | Seriousness to Subject if Risk Occurs |
| | None | | | |
| | Legal Risks: | Procedures to Protect Against / Minimize Risks | Likelihood of Occurrence | Seriousness to Subject if |
| | None | | | |
| , | Other Risks: | Procedures to Protect Against / Minimize Risks | Likelihood of Occurrence | Seriousness to Subject if Risk Occurs |
| | None | | | |
| 5.2 | | elated to the research activities<br>r payment, e.g. subject, sponso | | of standard of care and indicate who |
| Ba | accel Activity (includi | ng medication) Beyond Standa | rd of Caro | Party Responsible for Payment |
| ING. | Search Activity (motual | ing medication, beyond otanda | a or oare | There will be no additional expense incurred by the patient participating in this study. The patient's insurance carrier will be charged for anesthetic services received as per contract |
| j.3 | | osts that may be incurred by the or research related injury etc. I | | articipation in this study, e.g. travel |
| | itional Approvals for Di<br>ulations | rug Usage Required to Ensure | Risks are Minimiz | ed and Compliance with IND |
| 5.4 | | the use of drugs? (If no skip to | 5.11, if yes comple | ete 5.5 – 5.10.) X YES 🗆 No |
| 5.5 | attach 1) confirmation<br>Manufacturing Practic | from the manufacturer of com | ipliance with fede<br>he IND # is not pro | ly. For studies involving INDs also<br>ral regulations and Good<br>ovided, a letter from the sponsor |

| Drug Name | Dosage,<br>Frequency &<br>Duration | Method of<br>Administration | IND # if<br>Available | Manufacturer of IND | Sponsor<br>of IND | Supporting<br>Documents<br>Attached |
|---|---|---|---|---|---|---|
| Liposomal<br>Bupivacaine<br>(Exparel)<br>Experimental<br>Group | 0.4% 60ml<br>solution, once | Injection | n/a | n/a | l n/a | n/a |
| Bupivicaine<br>Control<br>Group | 0.25% 60ml<br>solution, once | Injection | n/a | n/a | n/a | n/a |

5.6 Provide the following Information relating to the storage, inventory and dispensing of drugs used in this study. Investigational drugs must be stored in the hospital Pharmacy unless the investigator ensures that storage, dispensing, accountability, and security comply with institutional policy and federal and state laws. The Director of Pharmacy, or delegated pharmacy staff, must approve plans for control of investigational drugs maintained outside of the pharmacy. Investigators who choose to store investigational drugs outside the Pharmacy will be subject to regular auditing by the Pharmacy.

Where will drugs be stored? Anesthesia carts

Describe the storage area and how it meets the required storage conditions for the drug: Anesthesia carts within the Ambulatory Surgery Center

Describe the security measures in place for inventory control and monitoring of the drug inventory: Locked carts

How and by whom will drugs be dispensed? Anesthesiologist performing the procedure

Describe how the disposition of unused drugs will be handled: Unused drugs and syringes are disposed in locked sharps boxes

Drug costs, when applicable, and other Pharmacy expenses associated with the study will be charged to the investigator and must be properly allocated for in the research contract or study budget and reimbursed to the Pharmacy. A department budget or special fund account will need to be provided to the Pharmacy from which the following fees will be drawn: N/A

- 1. Study initiation (one time fee)
- 2. Randomization (per subject enrolled)
- 3. Drug preparation and dispensing (per dose)
- 4. Drug cost (for non-sponsored studies)
- 5. Inventory and record keeping (monthly fee which includes quality assurance measures, monitor site visits, and drug storage)
- 6. Study closure (one time fee which includes destruction of remaining drug, copying and archiving study related information)
- \*Note that even if the Pharmacy is not storing or dispensing study drugs, study initiation fees will be charged to cover the costs of protocol review and to ensure that drugs not handled by the Pharmacy are in accordance with regulatory standards.

Additional Information Regarding an Investigational New Drug Application. (If yes to 5.8, 5.9 or 5.10 an IND is needed).

- 5.7 Has an IND already been obtained for the drug(s) used within the study? (If no, answer 5.8 5.10. If yes, be sure information requested in 5.5 is provided and skip to 5.11) 

  YES X No
- 5.8 Is the proposed investigation intended to be reported to the FDA in support of a new indication or to support any other significant change in the labeling for the drug? ☐ YES X NO

| Is the investigation intended to support a significant change in the advertising for the product? ☐ YES X NO | | | | | |
|---|---|---|---|---|---|
| other factor that sig | inificantly inc | reases the risks | s (or decreases t | | |
| itional Information fo | r Investigation | nal Devices | | · ·· | |
| Will the study invol | ve the use of | an investigation | nal device? (if no | skip to 5.15, if yes com | nplete 5.12 -5.14) |
| the manufacturer of | f compliance v | manufacturer. F<br>with federal reg | or studies involutions and Go | ving IDEs also attac<br>ood Manufacturing F | th confirmation from<br>Practices and of IDE |
| Device Name | IDE Number | | | Confirmation of | Confirmation of IDE |
| | | of IDE | of IDE | GMP Attached | Approval Attached |
| For NSR devices, at device, the propose procedures. The sp | ttach the spored investigation on the contract of the contract | nsor's descript<br>onal plan, a des<br>also inform the | ion of the device<br>cription of patie | e, reports of prior in<br>nt selection criteria | vestigations with the and monitoring |
| Describe plans for | maintaining i | nventory of the | investigational | device. | |
| Where will the devic | e be stored? | | | · | |
| Describe measures | in place for in | ventory contro | l: | | |
| Describe measures | for monitorin | g / tracking of t | he device: | | |
| How and by whom v | vill the device | be used? | | | |
| Describe plans for r | eturn of unus | ed devices to t | he sponsor: | | |
| itional Approvals Red | quired from ti | he Institutional | Biosafety Comm | | |
| If ves provide proof | f of approval f | for the study fr | om the Institutio | nal Biosafety Com | mittee. (Approval from the ecombinant DNA.) |
| TION 6 -REASONABLEN | ESS OF RISKS IN | N RELATION TO B | ENEFITS, IF ANY (4 | 5 CFR 46.111(A)(2)) | |
| | | | | ne PI, is associated | with this study. |
| Risk Level | | X to select | Comments | | |
| None | | | | | 1 |
| Minimal | u Ballutur - 1 | | | | |
| Minimal Slight Increase Ove | r Minimal | X | | | |
| | Does the investigat other factor that sig with the use of the ditional Information for Will the study involed YES X NO Provide Name, IDE the manufacturer of approval from the series Device Name Is the device consister NSR devices, and device, the propose procedures. The sign what determination Describe plans for Where will the device Describe measures Describe measures How and by whom who who will be plans for respect to the project in lifty yes provide procedures the project in lifty yes provide | Does the investigation involve a other factor that significantly inc with the use of the drug product with the use of the drug product with the use of the drug product with the use of the drug product with the use of the drug product will the study involve the use of YES X NO Provide Name, IDE number and a the manufacturer of compliance approval from the sponsor. Device Name IDE Number Is the device considered a significant for NSR devices, attach the spondevice, the proposed investigation procedures. The sponsor must a what determination was made by Describe plans for maintaining in Where will the device be stored? Describe measures in place for in Describe measures for monitorin How and by whom will the device Describe plans for return of unusual institutional Biosafety Committee must be considered and X after the level of over Comments may also be provided to Risk Level | Does the Investigation involve a route of adminiother factor that significantly increases the risks with the use of the drug product? YES X No litional Information for Investigational Devices Will the study involve the use of an investigation YES X No Provide Name, IDE number and manufacturer. Fithe manufacturer of compliance with federal regapproval from the sponsor. Device Name IDE Number Manufacture of IDE Is the device considered a significant risk or no For NSR devices, attach the sponsor's description device, the proposed investigational plan, a desprocedures. The sponsor must also inform the what determination was made by those IRBs. Describe plans for maintaining inventory of the Where will the device be stored? Describe measures in place for inventory control Describe measures for monitoring / tracking of the How and by whom will the device be used? Describe plans for return of unused devices to the Inventor of the Stitional Approvals Required from the Institutional Does the project involve the use of recombinant if yes provide proof of approval for the study from the Institutional Biosafety Committee must be obtained prior to see Tion 6 – REASONABLENESS OF RISKS IN RELATION TO Berick Place an X after the level of overall risk that, in Comments may also be provided to justify the assertion of the Institution of the Institution of the Institution of Institution of the Institution of Instituti | Does the Investigation involve a route of administration or dosa other factor that significantly increases the risks (or decreases twith the use of the drug product? YES XNO itional Information for Investigational Devices Will the study involve the use of an investigational device? (If no YES XNO Provide Name, IDE number and manufacturer. For studies involve the manufacturer of compliance with federal regulations and Go approval from the sponsor. Device Name IDE Number Manufacturer Sponsor of IDE Is the device considered a significant risk or non-significant risk For NSR devices, attach the sponsor's description of the device device, the proposed investigational plan, a description of patie procedures. The sponsor must also inform the IRB if other IRB what determination was made by those IRBs. Describe plans for maintaining inventory of the investigational Where will the device be stored? Describe measures in place for inventory control: Describe measures for monitoring / tracking of the device: How and by whom will the device be used? Describe plans for return of unused devices to the sponsor: Itional Approvals Required from the Institutional Biosafety Committee must be obtained prior to seeking IRB approval for TION 6—REASONABLENESS OF RISKS IN RELATION TO BENEFITS, IF ANY (4 Place an X after the level of overall risk that, in the opinion of the Comments may also be provided to justify the assessed risk level. | Does the Investigation involve a route of administration or dosage level, or use in a other factor that significantly increases the risks (or decreases the acceptability of with the use of the drug product? |

| 6.1 | What benefit, if any, may be gained by the subject and/or society? Discuss why the risks to subjects are reasonable in relation to the anticipated benefits to subjects and others. Participation in this study will not directly benefit patients, except that the injection of liposomal bupivacaine may provide longer duration of pain control after surgery than the injection of bupivacaine. It will improve our understanding of the efficacy of injecting long acting local anesthetic infiltration analgesia in managing postoperative analgesia in hip arthroscopy patients |
|---|---|
|---|---|

- Discuss the importance of the knowledge that may be gained as a result of the proposed research.

  Discuss why the risks to subjects are reasonable in relation to the importance of the knowledge that may result. The knowledge gained from this research may provide a method of longer pain control with fewer side effects and earlier mobilization of patients. In the unlikely case that patients receiving local infiltration analgesia may experience more pain, they will be able to receive pain medications without any restriction to keep them comfortable. We expect that both the experimental and control arms of the study will provide better analgesia with fewer side effects when compared to conventional use of narcotic pain medications.
- 6.3 For studies requiring full board review, describe the scientific review process that the study has undergone. Reviewed by members of Anesthesia Staff

SECTION 7 - SUBJECT SELECTION / RECRUITMENT DATA (45 CFR 46.111(a)(3) &(a)(7)(b))

7.0 Place an x after the type(s) of human subjects that are likely to be recruited for this study. SFHMC does not review/approve research involving prisoners.

| Pregnant Women or Fetuses | Children/Adolescents | Inpatients |
|---|---|---|
| Decisionally Impaired (for non-interventional studies only) | Viable Neonates | Outpatients X |
| SFMHC Employees | Educationally Disadvantaged | Terminally III |
| Students, Residents, or Fellows | Economically Disadvantaged | Physically Disabled |
| Other (describe) | | |

Provide any additional comments to describe subject populations:

- 7.1 Explain why the inclusion of any vulnerable populations identified in 7.0 is necessary (vulnerable populations include pregnant women or fetuses, neonates, and children): N/A
- 7.2 What is the maximum number of subjects to be enrolled at SFHMC? 36 subjects
- 7.3 Explain on what basis it is reasonable to expect that recruitment goals will be met. We perform 100 hip arthroscopies a year at St. Francis Hospital and Medical Center
- 7.4 If applicable what is the national expectation for enrollment? N/A

Data Collection and Recruitment Methods

7.5 Place an x after the source(s) from which information will be collected.

| Medical interventions | X | Labs results | x |
|---|---|---|---|
| Existing directly identifiable specimens | | Identifiable Waste material | |
| Existing coded specimens | | De-identified Waste material | |
| Existing de-identified specimens | | Excess material | |
| Interviews | X | Medical records | - X |

| | Focus groups | | Research registry * | |
|---|---|---|---|---|
| Other sources of informat | tion (provide de | ecription): | - | |
| Other sources of informat | ion (provide de | sscription). | 1 2000 M 10 | |
| *Provide the name and IRI | B number of th | e registry that w | ill be used: | |
| | | | H = TE | |
| recruitment strategies | s will be imple<br>ns of recorded ads f | mented. (Note: Al | e used to recruit subjects and materials for and methods of recruitmen ovided. It is acceptable to identify a recru | t must receive IRB approval pric |
| Methods/Materials | X to Select | Description of | Implementation | |
| Radio spots | | | | |
| Newspapers | | | | |
| Magazines | | | | 2000 |
| Broadcast messages | | | | |
| Purchased mailing lists | | | | |
| Patient base | X | | | |
| Flyers | | 7 EZ | | |
| Phone Calls | | | | |
| Web postings | | | | |
| illowing elements: title: purpos | e of the study; pro | otocol summary; ba<br>oval must be sough | not require IRB approval when the paid of the light of the local of th | ion(s); and how to contact t |
| | al or other com | | vill be paid to the subjects and | i the disbursement |
| None | | | | |
| None Section 8 - Informed Consi | ENT PROCESS (4 | 5 CFR 46.111(A) | 4)) | |
| SECTION 8 – INFORMED CONSI | exempt status If no and study | or a waiver of the | 4)) e requirement to obtain consolliment, or you have requested exec | ent ? ☐ YES X No<br>mpt status and will be |
| BECTION 8 – INFORMED CONSI<br>B.0 Have you requested (<br>(If yes, skip to section 10 consenting subjects, com | exempt status If no and study plete all items in reference of co | or a waiver of the is open to new enrithis section.) | e requirement to obtain conse | mpt status and will be |
| BECTION 8 – INFORMED CONSI B.0 Have you requested (If yes, skip to section 10 consenting subjects, com B.1 Provide the version reinformed consent che | exempt status If no and study plete all items in reference of co ecklist. | or a waiver of the is open to new enrithis section. ) nsent form sub- | e requirement to obtain consections of the consection of you have requested exection of the consection | mpt status and will be |
| SECTION 8 – INFORMED CONSI 3.0 Have you requested ( (If yes, skip to section 10 consenting subjects, com 3.1 Provide the version r informed consent che | exempt status If no and study plete all items in reference of co ecklist. | or a waiver of the is open to new enrithis section. ) nsent form sub- | e requirement to obtain consections of the consection of you have requested exection of the consection | mpt status and will be |
| SECTION 8 – INFORMED CONSI 3.0 Have you requested of (If yes, skip to section 10 consenting subjects, com 3.1 Provide the version reinformed consent che 3.2 Who will be authorized. | exempt status If no and study plete all items in reference of co ecklist. | or a waiver of the is open to new enrothis section. ) nsent form sub- | e requirement to obtain consections of the consection of you have requested exemple of the consection | mpt status and will be |
| SECTION 8 – INFORMED CONSI 3.0 Have you requested (If yes, skip to section 10 consenting subjects, com 3.1 Provide the version reinformed consent che 3.2 Who will be authorized Name of individual(s) auti | exempt status If no and study plete all items in reference of co ecklist. | or a waiver of the is open to new enrothis section. ) nsent form sub- | e requirement to obtain consoliment, or you have requested exemitted for review and approval thorization? | mpt status and will be |
| SECTION 8 – INFORMED CONSI 3.0 Have you requested of (If yes, skip to section 10 consenting subjects, com 3.1 Provide the version reinformed consent che 3.2 Who will be authorized Name of Individual(s) authorized Sanjay Sinha | exempt status If no and study reference of co ecklist. ed to obtain co horized: | or a waiver of the is open to new enrothis section. ) nsent form substitutions of the image is a section of the image is | e requirement to obtain consections of the consection of the conse | mpt status and will be |

| 8.4 | Who will provide consent/permission (e.g. the subject, parent, LAR)? Note: LARs can consent only for non-interventional studies. Subject |
|---|---|
| 8.5 | If consent will be obtained from LARs, describe the process for ensuring that the LAR is in fact the court-<br>appointed conservator or guardian, or individual designated as having power of attorney for health care,<br>or individuals designated as a health care representative. Consent from next-of-kin is not acceptable<br>absent one of the prior designations. Note: LARs can consent only for non-interventional studies. |
| 8.6 | Will anyone other than the subject/LAR be a part of the consent process (e.g. witness)? ☐ YES X NO |
| 8.7 | How will the privacy of the subjects/LARs be maintained throughout the consent process? The patient will be consented in a private area prior to surgery. Study records and identities will be kept confidential. If the results of the study are published in a scientific journal or presented at a scientific meeting, the subjects names' and identifying information will not be disclosed. |
| | Describe in detail the process for obtaining consent, including steps that will occur, the estimated length of the discussion, and how will it be ensured that subjects / LARs have had enough time to consider their decision regarding participation. Note: the consenting process needs to be documented in the research record for each subject. During the preoperative evaluation, appropriate subjects will be asked to participate in the study. The procedures, risks, and benefits will be explained by at least one of the investigators. |
| 8.9 | How will on-going consent of the subjects /LARs be obtained throughout the conduct of the study? N/A |
| 8.10 | Will any screening activity occur prior to consent / authorization being obtained? ☐ YES X No |
| 8.1 | 1 Describe the process of obtaining assent from children or decisionally impaired adults. N/A |
| | 2 Provide any additional comments regarding the consent process. |
| Fn | suring There Is No Undue Influence Within the Consent Process |
| 8.1 | 3 Describe plans to minimize the possibility of coercion or undue influence during the consent process: Patients will be informed that they do not have to participate in the study; they will receive the same standard of care. Patients have the right to withdraw from the study anytime |
| 8.1 | 4 What benefit, if any, is to be gained by the research personnel for subject recruitment into the study, e.g. payment for enrollment? If applicable, disclose the value of the benefit and explain how it is justified. None |
| SE | CTION 9- INFORMED CONSENT DOCUMENTATION (45 CFR 46.111(A)(5) AND .117(C)) |
| 9.0 | X YES NO |
| 9. | Would the consent form be the only record linking the subject to the research study? X YES ☐ NO |
| 9.5 | The state of the s |
| 9. | If no, explain the rationale for this assessment. |
| 9. | 4 Does the research involve any procedures for which written consent is normally required outside of the research context? ☐ YES X No |

#### SECTION 10 - PROTECTION OF PRIVACY OF SUBJECTS & CONFIDENTIALITY OF DATA (45 CFR 46.111(A)(7) & HIPAA)

- 10.0 How will the privacy interest of subjects be maintained throughout the conduct of the study (note, privacy pertains to the individual not to the data)? Patients will be assigned a study subject number that will be used on all data collection documents. Their personal information (Name, address, telephone number, age, weight, height, sex, etc.) will only be recorded on one list with study subject numbers. This list will be separate from all other documents under lock and key and only used to make follow up phone calls. Study records are kept confidential. If the results of the study are published in a scientific journal or presented at a scientific meeting, the subjects' names and any identifiers will not be used.
- 10.1 What information, if any, will be sought from the subject about other living individuals? None

10.2 Describe the procedures to protect the confidentiality of data during the conduct of the study by addressing each element noted below (note, confidentiality pertains to the data, not the individual).

Who will own the data (Sponsor, SFHMC or the PI)? SFHMC

Describe plans for storage and security of information on hard copy, including how research records will be labeled and if applicable, how information will be protected during transportation from external sites and from SFHMC. Locked file cabinet in anesthesia office

Will lab results be posted to medical records or research records? Medical records

Will other study related information, e.g. the informed consent document, survey tools, be posted to the medical record or research record? Consent form and survey/data collection form will be placed in research record.

Describe plans for storage and security of identifiable/coded samples. N/A

Describe plans for storage and security of electronic data.

Password protected on a SFHMC computer

Describe the security measures that are in place for the equipment that houses identifiable data. Locked file cabinet

Who will have access to hardcopy, samples, and / or electronic data?

Pl. co-investigators, and coordinator

How will access be managed?

Under lock and key

Describe the plans for storage or destruction of identifiable data for screened failures.

Locked cabinet

10.3 Describe procedures to continue to protect confidentiality after study closure by addressing each element noted below.

How long will information continue to be stored? 1 year after study is closed, and then information will be archived at Iron Mountain for long-term storage (at least 5 years).

Describe plans for on-going storage and security of hard copy data. Lock and key, password protected

Describe plans for on-going storage and security of identifiable samples. None

Describe plans for on-going storage and security of electronic records. Password protected

Who will have access to hardcopy, samples and/or electronic data? PI, co-investigators, coordinator

How will access be managed? Under lock and key

Describe the plans for the destruction of identifiable data. Shredder

| CTION 11 -SAFETY MONITORING (45 CFR 46.111(A) | (6)) | | St. the temptal of and | -4.2 |
|---|---|---|---|---|
| O Place an X after the entity responsible for s<br>monitoring in place for this study. For mul<br>monitoring plan; and when applicable the I<br>meeting etc., and when possible summarie | ti-center trials, (<br>SMR charter d | or triais with extern<br>escribing details of | membership, frequen | cy of |
| ntity responsible for monitoring: | | If applicable descri | be other entities below. | <u> </u> |
| Monitoring internal to SFHMC:<br>Wesley Knauft, MD<br>Woodland Anesthesia<br>860-714-6654 | n/a | | | |
| Monitoring by sponsor | n/a | liiwii = | | |
| Monitoring by other entity (describe) | n/a | | | |
| Tonew asset | | | | |
| Data Safety Plan | Independe | Surphy Services | V III WILLY | |
| Data Safety Board | Other (des | cribe) | | 10 |
| <ul> <li>1.1 Describe plans for communicating signification impact the subject's willingness to continuous subjects. Subjects will receive a letter if the subjects.</li> <li>1.2 Provide a brief description of the resource accessibility/availability of such resources.</li> <li>Resource</li> </ul> | es available to description | or that relate to the ificant findings. conduct this study, a of resource is not | including the | |
| | resource | of Anesthesiology | Readily available | L_<br>R_ 0 |
| Financial resources (internal and external | | | | |
| Staff (e.g. for medical/professional intervention) | Nurses | gists, Surgeons, | Readily available | |
| I IIIGI VOIIGOIII | | | | |
| Equipment (e.g. crash carts, shielding, resuscitation equipment, etc.) | | earts, Crash carts,<br>n equipment | Readily available | |

| resource | /Availability |
|---|---|
| Department of Anesthesiology | Readily available |
| Anesthesiologists, Surgeons,<br>Nurses | Readily available |
| Anesthesia carts, Crash carts, Resuscitation equipment | Readily available |
| OR, PACU supplies | Readily available |
| n/a | n/a |
| Hospital | Hospital availability |
| Hospital based | Hospital availability |
| | Department of Anesthesiology Anesthesiologists, Surgeons, Nurses Anesthesia carts, Crash carts, Resuscitation equipment OR, PACU supplies n/a Hospital |

SECTION 12- ADDITIONAL INFORMATION PERTAINING TO GENETIC RESEARCH

12.0 Does the study involve genetic research? 

YES X No
If no skip to section 13. If yes, respond to the remaining questions in this section.

| 4 | 12.1 | Will findings related to the study be disclosed to the subject? YES X NO (If yes, answer 12.2 – 12.7. If no, skip to 12.8. Note that if the researchers plan to release findings the subjects must also be given the opportunity to decline receiving information.) |
|---|---|---|
| | 12.2 | Describe what information will be provided. |
| 30 | 12.3 | Describe who will provide the information to the subject. |
| | 12.4 | Describe at what point in the study the information will be provided. |
| 12.5 Describe by what means it will be provided. | | |
| ľ | 12.6 | Describe the reliability of information provided. |
| ŀ | 12.7 | Explain the basis upon which the disclosure decision was made. |
| | 12:8 | Will unexpected and/or unrelated findings be disclosed? Subjects will receive a letter if there are any significant findings |
| | 12.9 | If findings will be published, explain how the subject's confidentiality will be ensured. The subjects' names and any identifying information will not be used. |
| | | ON-13 — SIGNATURE OF PRINCIPAL INVESTIGATOR AND DATE |
| | | Indicate if this protocol, or one similar to it, has previously been denied approval by any IRB panel. If it has previously been denied approval, also provide details regarding the IRB that denied approval, for what reasons approval was denied, when it was denied and how the concerns have been addressed. |
| | r<br>t<br>c<br>S<br>E | Signature of Principal Investigator. The undersigned assures that all key study personnel 1) have completed the required human subjects training, 2) are knowledgeable of the protocol and the institutions policy for reporting manticipated problems, non-compliance (protocol deviations/violations) and adverse events, 3) commit to conducting the study in accordance with the protocol as approved by the IRB, state law, federal regulations, SFHMC policies and with the ethical principles of respect for persons, beneficence and justice as set forth in the selmont Report. The undersigned also accepts primary responsibility for all aspects of the management of this study. Date 06/10/13 |
| Si | gnati | ure |

| 1. ; |
|------|